CLINICAL TRIAL: NCT06232811
Title: Mother-to-infant Bonding and Prematurity Are Associated With Sensory Processing at 12 Months of Age
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Gazi University, Gazi University
Other Study IDs: E-77082166-604.01.02-639350
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Preterm; Sensory Disorder; Attachment Disorder
MeSH Terms: conditions — Premature Birth; Sensation Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm: preterm infants with gestational age <34 weeks
  Interventions: Behavioral: Assessment
- Term: term infants with gestational age >37 weeks
  Interventions: Behavioral: Assessment

INTERVENTIONS:
Behavioral: Assessment — Sensory processing skills of children in the preterm and term groups will be evaluated. Additionally, the attachment between mother and baby will be evaluated.

SUMMARY:
Establishing a strong bond between mother and infant is crucial for fostering healthy relationships in the future. This research sought to investigate the correlation between mother-to-infant bonding and sensory processing, as well as the connection between prematurity and sensory processing in 12-month-old infants.

DETAILED DESCRIPTION:
At the age of four months, mothers will utilize the Mother-Infant Attachment Scale (MIBS) to evaluate the bonding between themselves and their infants. Subsequently, at 12 months old, the sensory processing abilities of the infants will be assessed using the Test of Sensory Functions in Infants (TSFI). The study will encompass both preterm and term-born children.

ELIGIBILITY:
Inclusion Criteria:

preterm children with a gestational age <34 weeks Term children with a gestational age between 37 and 41 weeks

Exclusion Criteria:

* infants with chromosomal defects, metabolic or neuromuscular disease,
* hydrocephalus, cerebral palsy, congenital heart disease,

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm and term children aged 12 months
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Mother-to-Infant Bonding Scale | 15 minutes
  The Mother-to-Infant Bonding Scale is a tool designed for evaluating mother-infant bonding. Comprising 10 items on a 4-point scale, this scale yields a total score ranging from 0 to 30. Higher scores on the scale are indicative of poorer mother-to-infant bonding.
Test of Sensory Functions in Infants | 30 minutes
  The test consists of 24 items divided into five subtests: sensory processing and reactivity. subtests include: deep pressure, adaptive motor functions, visual-tactile integration, ocular-motor control, and vestibular stimulation. By observing the baby's response, items are scored from negative to normal according to the criteria provided; Items are given 0, 1 or 2 points depending on the baby's reaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)